CLINICAL TRIAL: NCT04083807
Title: A Randomised Controlled Multicenter Single-blinded Phase III Study to Evaluate the Efficacy and Safety of TISSEEL Lyo Compared to Manual Compression as an Adjunct to Haemostasis During Vascular Surgery
Brief Title: Efficacy and Safety of TISSEEL Lyo Compared to Manual Compression as an Adjunct to Haemostasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BXU529732
Record Dates: First submitted 2019-08-23; First posted 2019-09-10 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Adjunct to Hemostasis During Vascular Surgery
Keywords: haemostasis; tissue glue; tissue sealing; Ilio-femoral bypass; Femoro-femoral bypass; Ilio-popliteal bypass; Femoro-popliteal bypass; Femoro-tibial vessel bypass; Arterio-arterial-bypass; Arteriovenous shunting for dialysis
MeSH Terms: interventions — Solvents; Thrombin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TISSEEL Lyo (Experimental): Applied once intra-operatively to the study suture line using the DUPLOJECT Fibrin Sealant Preparation and Application System.
  Interventions: Biological: TISSEEL Lyo
- Manual compression with surgical gauze pads (Active Comparator): Treated once intraoperatively with manual compression using surgical gauze pads at the study suture line.
  Interventions: Procedure: Manual compression with surgical gauze pads

INTERVENTIONS:
Biological: TISSEEL Lyo — The dose to be applied is governed by variables including the type of surgical intervention, the size of the affected area and the mode of intended application, and the number of applications.. The guideline for sealing surfaces is one package of Tisseel Lyo 2 ml (i.e. 1 ml sealer protein solution plus 1 ml thrombin solution) is sufficient for a surface of at least 10 cm2.
  Other Names: Fibrin sealant Vapor Heated, Solvent/Detergent-Treated, with 500 IU/mL Thrombin
  Arms: TISSEEL Lyo
Procedure: Manual compression with surgical gauze pads — Surgical 4x4 inches gauze pads
  Arms: Manual compression with surgical gauze pads

SUMMARY:
The primary objective of the study is to evaluate the efficacy of TISSEEL Lyo for haemostasis in patients receiving peripheral vascular prosthetic expanded polytetrafluoroethylene (ePTFE) conduits, as compared to a control arm treated with manual compression with surgical gauze pads.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* Male or female ≥ 18 ages;
* Patients undergoing primary vascular surgery (i.e., conduit placement with an ePTFE graft), including the following:

  1. Arterio-arterial-bypass;

     * Ilio-femoral bypass;
     * Femoro-femoral bypass;
     * Ilio-popliteal bypass;
     * Femoro-popliteal bypass;
     * Femoro-tibial vessel bypass
  2. Arteriovenous shunting for dialysis access in the upper or lower extremity;

Intraoperative inclusion criterion:

* Suture line bleeding eligible for study treatment is present after surgical hemostasis.

Exclusion Criteria:

* Concurrent participation in another clinical study treatment with another investigational drug or device within last 30 days;
* Other vascular procedures during the same surgical session;
* Arterio-arterial bypasses with more than two anastomoses;
* Haemoglobin <9.0 g/dL at screening;
* Pregnant or lactating women;
* Congenital or acquired coagulation disorders;
* Prior kidney transplantation;
* Heparin-induced thrombocytopenia;
* Known prior exposure to aprotinin within the last 12 months;
* Known hypersensitivity to aprotinin, heparin, blood products or other components of the investigational product;
* Unwilling to receive blood products.
* Known severe congenital or acquired immunodeficiency;
* Prior radiation therapy to the operating field;
* Severe local inflammation at the operating field;
* Positive results of any of the following the blood tests: HIV, syphilis, hepatitis B, hepatitis C.
* Emergency surgery.
* Alcohol or drug abuse.

Intraoperative exclusion criteria:

* Major intraoperative complications that required resuscitation or deviation from the planned surgical procedure;
* Intraoperative change in planned surgical procedure, which resulted in patient no longer meeting preoperative inclusion criteria or having preoperative exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2019-10-22 (Actual)

PRIMARY OUTCOMES:
Number of participants achieving hemostasis at 4 minutes after treatment | Day 0 (4 minutes post-treatment to closure of surgical wound)
  Performed on suture line.

SECONDARY OUTCOMES:
Number of participants achieving hemostasis at 6 minutes after treatment | Day 0 (6 minutes post-treatment to closure of surgical wound)
  Performed on suture line.
Number of participants achieving hemostasis at 10 minutes after treatment | Day 0 (10 minutes post-treatment to closure of surgical wound)
  Performed on suture line.
Number of participants with intraoperative re-bleeding after hemostasis | Day 0 (intraoperative)
  Performed on suture line.
Number of participants with postoperative re-bleeding after hemostasis | Day 1 (postoperative)
  Performed on suture line. Requires surgical re-exploration.

CONTACTS AND LOCATIONS:
Locations (5):
- Russia (5):
  - Baxter Investigational Site, Moscow
  - Baxter Investigational Site, Novosibirsk
  - Baxter Investigational Site, Rostov-on-Don
  - Baxter Investigational Site, Ryazan
  - Baxter Investigational Site, Saint Petersburg